CLINICAL TRIAL: NCT04751253
Title: The Combined Effect Of Different Doses Of High-Intensity Laser And Traditional Exercise On Pain And Function In Patients With Chronic Knee Osteoarthritis
Brief Title: High Intensity Laser and Exercises in Knee OA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mona Mohamed Ibrahim, Assistant Professor, Cairo University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: HILT and Knee OA
Record Dates: First submitted 2021-01-31; First posted 2021-02-12 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Chronic Knee Osteoarthritis
Keywords: knee; osteoarthritis; HILT; exercise; pain; function
MeSH Terms: conditions — Osteoarthritis; Motor Activity; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1500 J + exercises (Active Comparator): consist of 17 patients, they will receive the application of HILT with intensity 1500 J plus exercises.
  Interventions: Device: High Intensity Laser Therapy
- 3000 J + exercises (Active Comparator): consist of 17 patients, they will receive the application of HILT with intensity 3000 J plus exercises.
  Interventions: Device: High Intensity Laser Therapy
- exercises + sham LASER (Sham Comparator): consist of 17 patients, they will apply exercises plus sham LASER.
  Interventions: Device: High Intensity Laser Therapy

INTERVENTIONS:
Device: High Intensity Laser Therapy — different doses of energies of high-intensity LASER on pain and functional activity in patients with chronic knee OA.

SUMMARY:
The purpose of the study is to compare the effect of different doses of energies of high-intensity LASER on pain and functional activity in patients with chronic knee OA.

DETAILED DESCRIPTION:
Adding HILT to the traditional physical therapy program may reduce pain and improve the functional status of the affected joints. This may provide clinicians with an understanding of the different treatment modalities that may improve the quality of life of patients suffering from chronic knee OA. Which may benefit a wide range of individuals affected by this chronic and widespread disease all over the world.

Although little is known about the efficacy or mechanism of action of what has been termed ''high-intensity laser therapy'' using Nd: YAG lasers it has become commercially available in veterinary practice and is being marketed for the treatment of musculoskeletal disease. clinical research specific to Nd: YAG high-intensity laser therapy is required, as it is being used with little supporting evidence.

As there was no evidence about the best protocol for the treatment of knee OA as each study was using different doses, different sites of application, different number of phases, frequency of sessions, and the interval between sessions that make it difficult to have the best results. Specifically, the dosage range in literature was ranged from 1250 to 3000 J as total energy transmitted during one treatment session. The current study is an attempt to answer the question of which dosage of the energy of high-intensity LASER is more effective on pain and functional activities in patients with chronic knee OA at the third degree of osteoarthritis as determined by (Kellgren/Lawrence grading system) as it was recommended that LASER is an ideal treatment for subjects in the later stages of OA .

ELIGIBILITY:
Inclusion Criteria:

1. All subjects diagnosed as third degree chronic knee OA as determined by (Kellgren/Lawrence grading system) (Kellgren and Lawrence, 1957).
2. Aged between 50- 70 years
3. Persistent pain ≥4 on the visual analog scale (VAS) for more than 3 months in one or both knees.
4. Body mass index (BMI) ≤30 kg/m2.
5. Self-reported disability due to knee pain with a score of at least 25 on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC).
6. All subjects who will participate in this study will read, sign and date an informed consent form which required by ethical committee of faculty of physical therapy, Cairo university

Exclusion Criteria:

Patients will be excluded if they have the following conditions:

* History of joint replacement.
* Symptoms or signs suggestive of another cause of knee pain.
* Rheumatoid arthritis.
* Steroid injection or knee surgery (previous six months).
* acute inflammation around knee joint.
* Underlying disease such as malignancy.
* Infection or systemic disease of musculoskeletal system

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2021-02-02 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale | 8 weeks
  pain intensity
The functional disability assessment | 8 weeks
  The Western Ontario and McMaster Universities Osteoarthritis Index